CLINICAL TRIAL: NCT03885518
Title: Painted Playgrounds: A Scalable Approach to Increasing Physical Activity and Motor Skills in Louisiana Preschool Aged Children. Aim 2: Assessments
Brief Title: Painted Playgrounds: Aim 2: Assessments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Blue Cross Blue Shield (Other)
Responsible Party: Principal Investigator, Amanda Staiano, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PBRC 2017-040
Record Dates: First submitted 2019-01-29; First posted 2019-03-21 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Participants attending the childcare centers randomized to this arm will receive the stencil activities after baseline assessments have been completed. We will follow-up with assessments after 6-8 weeks
  Interventions: Other: Playground Stencils
- Wait-List (Placebo Comparator): Participants attending the childcare centers randomized to this arm will receive the stencil activities approximately 8 weeks after enrolling, after baseline and follow-up assessments have been completed.
  Interventions: Other: Playground Stencils

INTERVENTIONS:
Other: Playground Stencils — The stencils (hopscotch, agility trail, foursquare, bullseye, etc.) will be painted on the playgrounds at each childcare center. A toolkit and training video will be distributed to staff at each center to aid in instructing the children on how to perform the tasks.

SUMMARY:
The Painted Playgrounds Aim 2 (Assessment) project will examine the effects of a stenciling intervention aimed at increasing physical activity and improving fundamental motor skill functioning of preschool aged children. 72 children from local licensed childcare centers will participate in individual assessments at baseline and follow-up 6-8 weeks later. Assessments include height/weight, surveys and wearing a physical activity monitor (accelerometer) for 7 days. A parent/legal guardian will provide consent for their child to participate and will also complete a brief survey about their child's lifestyle and habits.

ELIGIBILITY:
Inclusion Criteria:

* A child who attends a childcare center enrolled to Aim 1.
* A child who is ≥ 3 years and ≤ 6 years old
* Your child will continue to attend this same childcare center for the duration of the study.

Exclusion Criteria:

• Parent/legal guardian is unwilling to provide written informed consent

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maura Kepper, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Background] Webster EK, Kepper MM, Saha S, Beyl RA, Kracht CL, Romain JS, Staiano AE. Painted playgrounds for preschoolers' physical activity and fundamental motor skill improvement: a randomized controlled pilot trial of effectiveness. BMC Pediatr. 2023 Sep 9;23(1):455. doi: 10.1186/s12887-023-04260-2. PMID 37689622

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: The children attending childcare centers randomized to this arm will have their physical activity and motor skills assessed; observations will be completed at baseline and 6-8 weeks after stencil activities have been painted at their center.
- Control Group: The children attending childcare centers randomized to this arm will have their physical activity and motor skills assessed; these centers will NOT have the stencils and their observations will still be completed at baseline and 6-8 weeks after baseline.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 32 | 19
Completed | 22 | 17
Not Completed | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Contorol: The children attending childcare centers randomized to this arm will have their physical activity and motor skills assessed; observations will be completed at baseline and 6-8 weeks after stencil activities have been painted at their center.
- Total: Total of all reporting groups
Arm/Group | Intervention | Contorol | Total
Number analyzed (Participants) | 32 | 19 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 19 | 51
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 15 | 7 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 6 | 29
  White | 7 | 12 | 19
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Moderate to Vigorous Activity (MVPA) During Recess
Description: To test the effectiveness of a promising (cost-effective, easily scalable) playground stenciling intervention to increase physical activity, change in MVPA during recess will be measured using accelerometers. The main outcome variable will be percentage of recess time spent in MVPA, measured objectively using a physical activity monitor (i.e. accelerometer).
Time Frame: Baseline and follow-up (6 to 8 weeks after playground stenciling)
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Control: The children attending childcare centers randomized to this arm will have their physical activity and motor skills assessed; these centers will NOT have the stencils and their observations will still be completed at baseline and 6-8 weeks after baseline.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 32 | 19
percentage of time | 1.4 (3.7) | 6.2 (4.1)

2. Primary Outcome: Change in Fundamental Motor Skill Development
Description: The Test of Gross Motor Development, 3rd edition (TGMD-3) was utilized to assess fundamental motor skills. The test consists of a total of 13 skills which are designed to assess locomotor (6 skills) and ball (7 skills). Children complete two trials, and if they meet the specified performance criteria, they are scored a 1. If they fail to meet the criteria, they are scored a zero. Trials 1 and 2 are added to get the raw scores of locomotor and ball skill. For locomotor, this range is from 0-46; for ball skills, children can score from 0-54. Raw scores are then converted to scaled scores based on the TGMD-3 age and gender charts. The scaled scores are added to determine a total scaled score. The total scaled score has a percentile ranking to determine what percentile the child is in (<1,>99). The post-TGMD-3 total percentile was subtracted for the change score from the baseline percentile. A positive value indicates an improvement in fundamental motor skills, where
Time Frame: Baseline and follow-up (6 to 8 weeks after playground stenciling)
Measure: Mean (Standard Deviation); unit: percentile
Groups:
- Intervention: The children attending childcare centers randomized to this arm will have their physical activity and motor skills assessed; observations will be completed at baseline and 6-8 weeks after stencil activities have been painted at their center.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 32 | 19
percentile
  Baseline | 21.2 (3.7) | 25.8 (4.8)
  Follow-up | 37.7 (4.4) | 34.1 (6.1)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/19
Other Adverse Events (participants affected / at risk) | 0/32 | 0/19

LIMITATIONS AND CAVEATS:
Limitations include the small sample for this pilot study. Only four schools were examined in one region of the United States, so results may only be generalizable to this area or to programs with similar characteristics. The limited access to concrete space in most ECE centers is a limitation that must be considered for the expansion of this intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT03885518/Prot_SAP_000.pdf